CLINICAL TRIAL: NCT02510690
Title: Factors Associated With Poor Dengue Outcomes in Malaysia
Status: Completed | Type: Observational
Sponsor: Clinical Research Centre, Malaysia (Other)
Collaborators: University of Malaya (Other)
Responsible Party: Principal Investigator, Dr. Goh Pik Pin, Doctor, Clinical Research Centre, Malaysia
Other Study IDs: NMRR-14-1275-22205
Record Dates: First submitted 2015-07-26; First posted 2015-07-29 (Estimated); Last update posted 2017-02-02 (Estimated); Status verified 2017-02

CONDITIONS: Dengue Fever
MeSH Terms: conditions — Dengue

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This study aims to analyse the results of national data collected by the e-Dengue Information System in order to determine the factors associated with disease outcomes in all patients registered from January 2013 to December 2014.

DETAILED DESCRIPTION:
Dengue is the most important arthropod borne viral disease in humans. The World Health Organization has estimated that more than 70% of the global at risk population live in the WHO southeast Asia and Western Pacific region, which account for nearly 75% of global disease burden from dengue. The number of reported cases of dengue in Malaysia has increased fourfold from 44.3 per 100 000 population in 1999 to 181 per 100 000 in 2007. Serologically confirmed cases are approximately half of the number of reported cases. An increase in dengue deaths in the adult populations has been observed since 2002. A study in Vietnam showed that women and children appear to have increased risk of dengue shock syndrome and death. Children aged 6-10 years had highest risk of Dengue Shock Syndrome (DSS). However, mortality was highest in younger children. However, in a study of 560 adult dengue patients in Martinique, Thomas L et al found that severe dengue were mainly in males, elderly, and presented with abdominal pain, cough and diarrhoea. At present, there is no vaccine or cure for dengue. Treatment is mainly supportive and for symptom relief. Various measures have been employed to decrease the incidence of dengue - these have been mainly by public health measures. However, 2014 has seen a dramatic rise in the number of confirmed dengue cases as well as mortality.

This study aims to analyse the results of national data collected by the e-Dengue Information System in order to determine the factors associated with disease outcomes in all patients registered from January 2013 to December 2014.

An epidemiological observational study will be done by utilizing e-dengue data from year 2013 till year 2014. The inclusion criteria is all dengue cases registered in the e-Dengue information system 2013-2014; and there is no exclusion criteria.

The primary outcome measurement is the disease outcome which included recovery, hospitalisation and death.

All data collected will be analyzed by using descriptive analysis, the prevalence/incidence will be estimated; and regression model will be generated.

ELIGIBILITY:
Inclusion Criteria:

* All dengue cases e-Dengue Information System 2013-2014

Exclusion Criteria:

* Nil

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All dengue cases that registered under e-Dengue Information System 2013-2014
Sampling Method: Non-Probability Sample
Enrollment: 20000 (Actual)
Dates: Start 2014-10; Primary Completion 2016-01 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Mortality rate | through out the length of hospital stay, an average of 7 days
  to determine the mortality rate secondary to dengue
The proportion of dengue patient who recover from dengue and discharged | through out the length of hospital stay, an average of 7 days
Number of participants with Disease severity | through out the length of hospital stay, an average of 7 days
  according to WHO classification

CONTACTS AND LOCATIONS:
Locations (1):
- Clinical Research Centre, Hospital Kuala Lumpur, KualaLumpur, Malaysia